CLINICAL TRIAL: NCT02526134
Title: Placing Trust in Endoscopic Ultrasonography: Impact on Planning Conformal Radiotherapy of Cancer of the Esophagus and Rectum
Acronym: FIDUCOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Cook medical laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIDUCOR-IPC 2013-008
Record Dates: First submitted 2015-06-25; First posted 2015-08-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-02

CONDITIONS: Oesophageal Cancer; Rectal Cancer
Keywords: Laying of medical devices (radio opaque markers)
MeSH Terms: conditions — Esophageal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laying of medical devices (Experimental): radio opaque markers
  Interventions: Device: radio opaque markers (Echo Tip Ultra Fiducial Needle - ETUF)

INTERVENTIONS:
Device: radio opaque markers (Echo Tip Ultra Fiducial Needle - ETUF)

SUMMARY:
The purpose of this study is to estimate the rate of patients in whom a significant change in the area to be irradiated will be observed between the assessment before and after laying the evaluation of Trustees.

DETAILED DESCRIPTION:
The centering of radiotherapy is done with the pre-radiation scanner for tracking the implementation of target skin markers. On this scanner, it is often difficult for the radiation therapist to pinpoint the target volume. To improve the definition of the target volume, image fusion techniques with other imaging tests were developed.

To improve the pre-radiotherapy identification, setting up markers echo-endoscopy has been described without major complications. The impact on targeting radiotherapy was mainly described for the prostate.

The marking of digestive tumors was described by the establishment of Trustees, radiopaque markers in the lymph nodes, esophagus, stomach, pancreas, and bile ducts.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Rectal cancer diagnosis or esophagus
* Radiotherapy indication
* Signed consent to participate
* Patient affiliated to a social security system or benefiting from such a system

Exclusion Criteria:

* Pregnant women, of child-bearing potential, or lactating women
* Patient deprived of liberty or under supervision of a guardian
* Impossibility to undergo medical examinations of the study for geographical, social or psychological reasons
* Contra-indication for procedure study (infeasible EUS)
* Contra-indication for general anesthesia
* Patient (e) with disorders of hemostasis
* Patient (e) with portal hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-04; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Patients rate in which a significant variation in the area to be irradiated will be observed between before evaluation and evaluation after laying the trustees. | From inclusion to 12 months follow up
  Observing whether there is a significant variation of the area to be irradiated

SECONDARY OUTCOMES:
Number of trustees (2 up 6 maximum) and set up their positions estimated success rate of implementation and the evaluation of the safety and toxicity (complications) associated with the establishment trustees (composite measure) | From inclusion to 12 months follow up
  Safety and security are measured by statistical analysis (numbers and percentage for qualitative variables and by average, median, standard deviations and extreme values for quantitative variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

REFERENCES:
- See also: official web site of the sponsor — http://www.institutpaolicalmettes.fr